CLINICAL TRIAL: NCT03018769
Title: Syndrome Differentiation in the Management of Chronic Stable Coronary Artery Disease (SCAD) to Improve Quality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Bi Yingfei, doctor, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Other Study IDs: FirstTeachingHTianjinUTCM
Record Dates: First submitted 2017-01-07; First posted 2017-01-12 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Stable Coronary Artery Disease
MeSH Terms: interventions — Ephedrae herba

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- chronic SCAD
  Interventions: Drug: Chinese Herb

INTERVENTIONS:
Drug: Chinese Herb

SUMMARY:
1.1 To build a TCM diagnosis and treatment database for chronic stable CAD; 1.2 To summarize the pattern of TCM medicine used and the effect of the medication in chronic stable CAD.

1.3 To formulate a syndrome differentiation determined medicine plan based on the improvement in the quality of life on chronic stable CAD patients.

DETAILED DESCRIPTION:
Chronic stable coronary artery disease (SCAD) is a general term for all kinds of coronary artery disease (CAD) which includes patients with chronic stable angina, oldmyocardial infarctions and also stable condition after revascularization (i.e percutaneous coronary intervention （PCI）, coronary artery bypass graft （CABG）). According to 2012 American Heart Association/American College of Cardiology (AHA/ACC) guide, the objective of the treatment for SCAD is to maintain or recover patients' exercise tolerance, quality of life and avoid complication like heart failure，so as to decrease mortality, eliminate symptoms and avoid adverse reactions.

Traditional Chinese medicine (TCM) has two thousand years of history in managing CAD and has its advantages in improving quality of life. Using scientific method to evaluate, demonstrate and conclude the clinical curative effect of TCM is an extremely important task for both TCM and Chinese and western integrative medicine win the treatment of CAD. Recent researches mainly focus on certain types or some certain pathological and physiological stages of CAD, worse still, different areas experts have their own experiences and opinions with the treatment. There is a lack of unified syndrome differentiation and prescriptions plan for the chronic stable CAD and not enough attention has been paid to TCM despite it having many advantages in improving quality of life in these patients. Considering all the above, this research studied past syndromes research results and real clinical effective chronic SCAD cases. Cases were analysed and explored, effective cases were filtered, syndrome differentiation of the prescriptions was refined, thus build a TCM diagnosis and treatment information database.

ELIGIBILITY:
Inclusion Criteria:

* without age limit
* diagnose as chronic SCAD at first visit
* heart function classification between II~III Canada classification(CCS)
* Be willing to accept Chinese herbal decoction
* sign an informed consent

Exclusion Criteria:

* suffer from acute myocardial infarction (AMI) ,unstable angina or prior revascularization(i.e PCI,CABG) in the latest 60 days .
* have such diseases as follow: a.poorly controlled blood pressure even taken medicine(systolic pressure≥180mmHg, diastolic pressure≥100mmHg); - severe arrhythmia(atrial fibrillation with rapid ventricular response, atrial flutter, paroxysmal ventricular tachycardia, etc); c.pulmonary heart disease, rheumatic heart disease, myocarditis, cardiomyopathy, aortic dissection, pulmonary embolism.
* hyperthyreosis, cervical spondylosis, gallbladder-cardiac syndrome, gastroesophageal reflux, esophageal hiatal hernia, neurosis, climacteric syndrome and other diseases which would cause chest pain.
* alanine transaminase(ALT) or serum creatinine(Scr) more than twice the normal reference value.
* hemoglobin(Hb)<100g/L or have severe hematological system disease.
* malignant tumor.
* pregnant, lactating women or other women have reproductive requirement.
* psychosis or cognition impairment person.
* taken chinese medicine decoction in recent two weeks.
* not take part in any other clinical trail.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: chronic stable Coronary Artery Disease
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
EuroQol-5 Dimensions (EQ-5D) | change from take chinese herb in one week
Four diagnostic method of TCM | change from take chinese herb in one week
electrocardiograms(ECG) | change from take chinese herb in one week
dynamic electrocardiogram | change from take chinese herb in one week
ultrasonic cardiogram | change from take chinese herb in one week
treadmill exercise testing (TET) | change from take chinese herb in one week

CONTACTS AND LOCATIONS:
Locations (32):
- China (32):
  - The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine, Anhui
  - Beijing Hospital of Traditional Chinese Medicine, Beijing
  - Dongfang Hospital of Beijing University of Chinese Medicine, Beijing
  - Dongzhimen Hospital Affiliated to Beijing University of Chinese Medicine, Beijing
  - Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing
  - the third Affiliated to Beijing University of Chinese Medicine, Beijing
  - Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing
  - Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun
  - Affiliated Hospital of Gansu University of Chinese Medicine, Gansu
  - Guangdong Provincial Hospital of Chinese Medicine, Guangdong
  - Guangdong Second Troditional Chinese Medicine Hospital, Guangdong
  - First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou
  - Heilongjiang Provincial Hospital of traditional Chinese Medicine, Heilongjiang
  - Henan Province Hospital of TCM, Henan
  - The First Affiliated Hospital of Henan University of TCM, Henan
  - Affiliated Hospital of Hunan Academy of Chinese Medicine, Hunan
  - The First Hospital of Hunan University of Chinese Medicine, Hunan
  - The Second Affiliated Traditional hospital of Hunan University of Traditional Chinese Medicine, Hunan
  - Jiangsu Province Hospital of TCM, Jiangsu
  - Jiangxi Provincial Hospital of Chinese Medicine, Jiangxi
  - Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Liaoning
  - The Second Affiliated Hospital of Liaoning University of traditional Chinese Medicine, Liaoning
  - Shandong Province Hospital of Traditional Chinese Medicine, Shandong
  - Shanxi Hospital of Traditional Chinese Medicine, Shanxi
  - Shanxi Province Hospital of Traditional Chinese Medicine, Shanxi
  - The Affiliated Hospital to Shanxi University of Traditional Chinese Medicine, Shanxi
  - The Second Affiliated Hospital of Shanxi University of Traditional Chinese Medcine, Shanxi
  - Shijiazhuang Traditional Chinese Medicine Hospita, Shijiazhuang
  - First Teaching Hospital of Tianjin University of TCM, Tianjin
  - Second Affiliated Hospital of Tianjin University of TCM, Tianjin
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin
  - Traditional Chinese Medicine Hospital of Xinjiang Uygur Autonomous Region, Xinjiang